CLINICAL TRIAL: NCT00460837
Title: Virtual Colonoscopy: Comparison of Reduced Laxative Virtual Colonoscopy Regimens With Standard Preparation on Patient Experience and Compliance - a Questionnaire Based Study
Brief Title: Comparison of Bowel Preparation in Virtual Colonoscopy (VC) - Patient Experience
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Supply of adequate label was not provided to the MHRA
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Dr Alan Warnes, North West London Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 07.senna.SMH
Record Dates: First submitted 2007-03-23; First posted 2007-04-17 (Estimated); Last update posted 2010-07-26 (Estimated); Status verified 2010-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; bowel preparation regimen; patients with symptoms attributable to colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 A (Active Comparator): gastrofin & Picolax
  Interventions: Drug: bowel preparation: senna & gastrofin versus picolax (standard)
- 2 (Active Comparator): senna
  Interventions: Drug: bowel preparation: senna & gastrofin versus picolax (standard)

INTERVENTIONS:
Drug: bowel preparation: senna & gastrofin versus picolax (standard) — The intervention is a bowel cleansing procedure

SUMMARY:
The study will compare patient's experience between those taking a standard bowel cleansing regimen with minimal laxative tagging regimen of senna and gastrofin. Additionally comparing any possible reduction in diagnostic accuracy that may ensue from an increased quantity of retained faecal residue.

DETAILED DESCRIPTION:
Bowel cleansing with high dose laxative is the standard bowel preparation prior to whole colon investigations but such regimens are associated with considerable patient discomfort and inconvenience, potentially affecting compliance rates [1-3].

Unlike existing whole colon investigations (conventional colonoscopy and barium enema), reduced laxative regimens can be successfully used with VC, with the aim of improving patient experience, whilst maintaining diagnostic accuracy. These regimens utilize faecal tagging; a method of labeling residual faeces and fluid with radiodense liquids, such as iodine or barium based fluids, which are taken orally by the patient. Once faecal residue and fluid is labeled in this way, it can easily be discriminated from true pathology (which remains 'untagged').

We are proposing to compare different bowel preparation regimens, and ascertain patient experience of the different regimes, while monitoring diagnostic accuracy of the 2 different regiments.

ELIGIBILITY:
Inclusion Criteria:

* patients with symptoms attributable to colorectal cancer

Exclusion Criteria:

* patients with known colorectal cancer referred for staging VC
* patients who take laxatives regularly or with previous inadequate colonic examination due to excessive faecal residue
* patients deemed too frail to undergo full bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-11; Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Versus standard bowel preparation | 1 day (while on regimen + effectivness analysis time)
Patient experience and compliance with reduced laxative tagging versus standard preparation | 1 day (while on regimen)

SECONDARY OUTCOMES:
Comparison of per polyp specificity between the two preparation regimens | 1 day (analysis time)

CONTACTS AND LOCATIONS:
Overall Officials: David Burling, Principal Investigator — St Mark's Hospital, North West London Hospitals NHS Trust
Locations (1):
- St Mark's Hospital, North West London Hospitals NHS Trust, London, Middlesex, United Kingdom